CLINICAL TRIAL: NCT00214695
Title: A Subjective Evaluation of Inflow Pain Associated With the Use of an Experimental Solution for Peritoneal Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRO-RENAL-REG-064
Record Dates: First submitted 2005-09-08; First posted 2005-09-22 (Estimated); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

INTERVENTIONS:
Drug: Experimental Peritoneal Dialysis Solution

SUMMARY:
The purpose of this study is to evaluate the inflow pain using an experimental peritoneal dialysis solution compared to a current solution for the management of end stage renal disease (ESRD) in peritoneal dialysis (PD) patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given written informed consent after the nature of the study has been explained.
* Patients who are at least 18 years of age.
* Patients who have been treated with PD using specific solutions for at least 30 days before the screening visit.
* Patients who experience pain on infusion based on medical judgement.

Exclusion Criteria:

* Patients who have received antibiotics for the treatment of an episode of peritonitis within 30 days before to screening visit.
* Patients who have had acute or chronic exit-site or tunnel infection in the past 14 days, counted from the last day of infection to the screening visit.
* Patients who are participating in another study that requires Ethics Committee approval. Non-interventional studies are permitted.
* Patients who have received an investigational product within 30 days preceding the screening visit.
* Patients who are pregnant or lactating. (NB: Female patients of childbearing potential must have a negative urine or serum pregnancy test at the time of the screening and will be required to use a medically acceptable means of contraception during their participation in this study).
* Patients who have a significant psychiatric disorder or mental disability that could interfere with his/her ability to provide informed consent and/or comply with protocol procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-05; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Locations (1):
- Huddinge Sjukhus, Njurmed kliniken K 56, Huddinge, Sweden